CLINICAL TRIAL: NCT03882866
Title: 3D-printed Template for Iodine-125 Seed Implantation Therapy in Patients With Locally Advanced Pancreatic Cancer: a Multicenter Study
Brief Title: Iodine-125 Seed Implantation Therapy for Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Hebei General Hospital (Other); Zhongda Hospital (Other); Anhui Provincial Hospital (Other Government); The Second Hospital of Shandong University (Other); Sun Yat-sen University (Other); Chinese PLA General Hospital (Other); Huadong Hospital (Other); Tengzhou Central People's Hospital (Other Government)
Responsible Party: Principal Investigator, Zhongmin Wang, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018clinicethicreview215
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: Iodine-125; Three-Dimensional Printing; Brachytherapy; template
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed non-coplanar template (Experimental): 3D-printed non-coplanar template is used in this group.
  Interventions: Procedure: 3D-printed non-coplanar template
- 3D-printed coplanar template (Active Comparator): 3D-printed coplanar template is used in this group.
  Interventions: Procedure: 3D-printed coplanar template

INTERVENTIONS:
Procedure: 3D-printed non-coplanar template — 3D-printed non-coplanar template is used in the intervention group. Iodine-125 seed implantation therapy is assisted using 3D-printed non-coplanar template as a guide in patients with locally advanced pancreatic cancer. 3D-printed non-coplanar template is designed and printed according to a preoperative CT scan and treatment planning system.
  Arms: 3D-printed non-coplanar template
Procedure: 3D-printed coplanar template — 3D-printed coplanar template is used in the intervention group. Iodine-125 seed implantation therapy is assisted using 3D-printed coplanar template as a guide in patients with locally advanced pancreatic cancer. 3D-printed coplanar template is designed and printed according to a preoperative CT scan and treatment planning system.
  Arms: 3D-printed coplanar template

SUMMARY:
This study evaluates the application of 3D-printed template for iodine-125 seed implantation therapy in patients with locally advanced pancreatic cancer. Half of participants will receive 3D-printed coplanar template, while the other half will receive 3D-printed non-coplanar template.

DETAILED DESCRIPTION:
Dosimetric verification was performed after implantation. Pre- and postoperative D90, V100, and V150 were calculated. The success rate of iodine-125 seed implantation, dosimetric parameters, objective response rate (ORR)，overall survival (OS)，toxicities and quality of life of two treatment regimens and complications were analyzed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Cytologically or histologically confirmed pancreatic adenocarcinoma
* Inoperable locally advanced pancreatic cancer based on American Joint Committee on Cancer (AJCC) staging system (8th ed) (without distant metastasis)
* Single tumor size≤ 6 cm
* Karnofsky performance score （KPS）≥60
* Estimated survival ≥3 months
* Without other several comorbidity
* Participants must have adequate organ function:

  * WBC≥3×109/L; HGB≥90g/dL; PLT≥50×109/L
  * Aspartate Transaminase (AST)/alanine aminotransferase ( ALT) ≤3 × institutional upper limit of normal
  * Albumin≥3g/dL
  * Total bilirubin ≤3mg/dL
  * PT≤3 × institutional upper limit of normal or INR≤2.3
  * Creatinine ≤1.5 × institutional upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with other malignant tumors
* History of other anti-cancer therapy, including surgery,radiation, ablation and so on
* Pregnant or lactating women
* Patients with Immunodeficiency disease
* Several heart disease, for example: New York Heart Association (NYHA) class III/IV congestive heart failure，active coronary heart disease and severe arrhythmia
* Uncontrolled hypertension
* Ongoing or active infection (>grade 2 based on National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) 4.0 edition)
* Active tuberculosis
* Chronic renal insufficiency
* Other organ failure
* History of organ transplantation
* History of severe mental illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  ORR is defined as the proportion of the subjects in the analysis population who have a complete response (CR) or partial response (PR). Responses are based on assessments per RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  OS is defined as the time from randomization to death due to any cause, or censored at date last known alive.
Incidence of treatment-emergent toxicities of two treatment regimens in patients | 24 months
  The toxicity criteria of the Radiation Therapy Oncology Group (RTOG) were applied to assess the acute and late adverse effects of irradiation.
Quality of life of two treatment regimens in patients | 24 months
  Quality of life will be evaluated using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ)C30 Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Wang, MD, Principal Investigator — Ruijin Hospital
Locations (8):
- China (8):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Zhongda Hospital, Nanjing, Jiangsu
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Teng Zhou Central People's Hospital, Zaozhuang, Shandong
  - Huadong Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No